CLINICAL TRIAL: NCT04161703
Title: Effect of Focused Ultrasound on Abdominal and Intrahepatic Fat in Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Taha, ASSISTANT PROFESSOR, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T REC/012/00451.
Record Dates: First submitted 2019-11-09; First posted 2019-11-13 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- focused ultrasound, diet and exercises (Experimental)
  Interventions: Procedure: focused ultrasound, diet and exercise
- diet and exercises (Experimental)
  Interventions: Procedure: diet and exercise

INTERVENTIONS:
Procedure: focused ultrasound, diet and exercise — Focused Ultra Sound using a device of Mabel6 DUO Ultra Cavitation Technology produced by DAEYANG MEDICAL CO., KOREA applied on the abdominal region which extending bilaterally from the line extending from mid-axilla to iliac crest, and above from center of diaphragm to the line extending between two iliac crests below.
  an aerobic exercise 3 to5 times/week for 12 weeks in the form of walking on treadmill for 30 minutes with moderate intensity a weight maintenance diet, which ranged from 1700 kcal to 2200 kcal/day, which was calculated in an individual basis for each subject according to his BMR, throughout the study period (12 weeks) to ensure that the reduction in the circumference was due to the treatment intervention rather than due to their weight reduction
  Arms: focused ultrasound, diet and exercises
Procedure: diet and exercise — weight maintenance diet, which ranged from 1700 kcal to 2200 kcal/day, which was calculated in an individual basis for each subject according to his BMR, throughout the study period (12 weeks) to ensure that the reduction in the circumference was due to the treatment intervention rather than due to their weight reduction. All subjects in both groups (A & B) followed an aerobic exercise 3 to5 times/week for 12 weeks in the form of walking on treadmill for 30 minutes with moderate intensity (moderate intensity = 12-14 according to Borg Scale). The beginning period will be 15 mints and increased gradually until reaching 30 mints per time.
  Arms: diet and exercises

SUMMARY:
In recent years, a number of modalities have become available for the noninvasive reduction of adipose tissue. One of those is high intensity focused ultra sound (HIFU). The study aimed to discover the effect of Focused Ultrasound on localized abdominal fat size in fatty liver patients.

Methods: In total, 40 participants with a body mass index (BMI) 30-40 kg/m2, whose age ranged between 30 and 45 years, mild to moderate fatty liver (Liver to Spleen ratio < 1), and with waist-hip ratio (WHR) greater than 0.8 for females and greater than 0.95 for males were included. The participants were randomly assigned to two groups, one group received focused ultrasound, diet, and exercises (the study group) and the other group received exercises, and diet only (the control group), respectively. Measures were abdominal subcutaneous fat volume, abdominal visceral fat volume, and liver to spleen ratio (L/S ratio) were measured at the beginning of the study and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

participants with a body mass index (BMI) 30-40 kg/m2, whose age ranged between 30 and 45 years, mild to moderate fatty liver (Liver to Spleen ratio < 1), and with waist hip ratio (WHR) greater than 0.8 for females and greater than 0.95 for males were included

Exclusion Criteria:

abdominal hernias, severe diabetes or autoimmune diseases; patients with osteoporosis, phlebitis and thrombophlebitis; patients with metallic sections, articular prosthesis, intrauterine devices or a pacemaker; pregnant women; patients with a reduced nervous sensibility or with neurological pathologies; patients with obliterating arteriopathies and patients with important inflammatory processes or neoplastic diseases

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Abdominal subcutaneous and visceral fats volume measured by Computed tomography. | three months
  The abdominal fat volume will be measured by a new advanced application which called "Synapse 3D Lung and Abdomen Analysis".

SECONDARY OUTCOMES:
Liver to Spleen ratio (L/S ratio) | three months
  measurement of liver attenuation in Hounsfield units (LA) by multidetector CT scans of the abdomen at the level of the T12 to L1 intervertebral space and was used to estimate fatty liver (low LA=high fatty liver). The LA was determined by calculating the mean Hounsfield units of 3 regions of interest in the parenchyma of the right lobe of the liver

OTHER OUTCOMES:
height in meters and waist to hip ratio (WHR), | three months

CONTACTS AND LOCATIONS:
Overall Officials: Mona M Taha, PhD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alaini, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taha MM, Aneis YM, Mohamady HM, S A A, Elsayed SH. Effect of focused ultrasound cavitation augmented with aerobic exercise on abdominal and intrahepatic fat in patients with non-alcoholic fatty liver disease: A randomized controlled trial. PLoS One. 2021 Apr 28;16(4):e0250337. doi: 10.1371/journal.pone.0250337. eCollection 2021. PMID 33909662